CLINICAL TRIAL: NCT01881945
Title: Validation of Tools Studying Respiratory Physiology and it Interaction With Swallowing and Cardiac Physiology.
Brief Title: Validation of Study in Respiratory Physiology and it Interactions
Acronym: ValApPhI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2008-A00273-52
Record Dates: First submitted 2013-05-24; First posted 2013-06-20 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Life Experiences; Respiratory Function; Cardiac Function
Keywords: Swallowing; Hyperventilation
MeSH Terms: conditions — Respiratory Aspiration; Hyperventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physiological measurments (Experimental)
  Interventions: Other: Non-invasive physiological signal recording on healthy volunteer

INTERVENTIONS:
Other: Non-invasive physiological signal recording on healthy volunteer

SUMMARY:
The aim of the study was to validate tools of physiological signal processing and interpretation on healthy human volunteers in order to improve the understanding in respiratory physiology and its interactions with heart function, and swallowing.

ELIGIBILITY:
Inclusion Criteria:

* healthy subject
* between 18 and 60 years old

Exclusion Criteria:

* patient
* person protected by the law

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Heart rate | one measure within two weeks of inclusion
  Heart rate is calculated on electrocardiograph
end tidal CO2 | one measure within two weeks of inclusion
  end tidal CO2 of each breath measured with an infrared CO2 analyzer
Non invasive arterial pressure | one measure within two weeks of inclusion
Non invasive stroke volume | one measure within two weeks of inclusion
  measured with impedance cardiography
Inspiratory and expiratory times | one measure within two weeks of inclusion
  obtained for each breath with flow signal
Tidal volume | one measure within two weeks of inclusion
  obtained for each breath with flow signal

CONTACTS AND LOCATIONS:
Overall Officials: BRIOT Raphael, MCU-PH, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Laboratoire TIMC-IMAG, La Tronche, France

REFERENCES:
- [Derived] Besleaga T, Blum M, Briot R, Vovc V, Moldovanu I, Calabrese P. Individuality of breathing during volitional moderate hyperventilation. Eur J Appl Physiol. 2016 Jan;116(1):217-25. doi: 10.1007/s00421-015-3260-3. Epub 2015 Sep 23. PMID 26400417